CLINICAL TRIAL: NCT05125848
Title: Clinical Evaluation of the CM-1500 During Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zynex Monitoring Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZMS-1500-2021-Dialysis
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Fluid Loss; Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hemodialysis Single Group Assignment (Experimental): All enrolled subjects will be connected to the CM-1500 for monitoring during their hemodialysis session
  Interventions: Device: CM-1500

INTERVENTIONS:
Device: CM-1500 — The CM-1500 is a U.S. FDA cleared non-invasive monitoring device that simultaneously monitors five (5) parameters of a patient's body. A combination of these parameters is represented by a single number known as the Relative Index value. This value is indicative of relative changes in fluid volume.

SUMMARY:
The study is a prospective, single-arm, non-randomized, non-blinded, non-controlled, non-significant risk, single center study enrolling up to 20 subjects consented to undergo a hemodialysis session as a part of their standard prescribed treatment plan. Subjects will consent to undergo non-invasive monitoring with the CM-1500 during three (3) separate sequential hemodialysis sessions.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Ability and willingness to comply with the study procedures and duration requirements, including connection of the device to the left wrist/hand and maintaining relatively motionless during the session
* 18 years of age or older
* Planned to undergo a minimum of three (3) hemodialysis sessions within the two (2) weeks following enrollment.

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Undergone an amputation of the left upper extremity
* Subjects with left arm hemodialysis access only
* Diagnosed with dextrocardia
* Subjects who have a pacemaker
* Subjects who have any other underlying condition that would inhibit completion of participation in the study, per Investigator opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tolins, MD, Principal Investigator — InterMed Consultants
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hemodialysis Single Group Assignment
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hemodialysis Single Group Assignment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Average Relative Index Value Following a Hemodialysis Procedure
Description: The primary objective is to characterize the average CM-1500 Relative Index (RI) following a hemodialysis procedure. The RI is an investigational value which utilizes proprietary algorithms to combine the changes of multiple measured parameters (utilizing a weighted summation of percent change values) which are indicative of relative changes in fluid volume in adult patients into a single value. The RI is a unitless value with no set minimum or maximum, where 100 is a patient's baseline. Based on the nature of the RI itself, a direct interpretation of a positive or negative outcome cannot be derived from the absolute value, instead it could be used to monitor trending of a patient's parameters relative to their baseline. The average RI after dialysis procedure was calculated by averaging all measured RI values for all subject sessions (3 sessions per subject, totaling 45 sessions) during the 10-min post-hemodialysis recovery period.
Time Frame: Duration of post-hemodialysis recovery period (10-minutes)
Measure: Mean (Standard Deviation); unit: Relative Index (RI)
Groups:
- Hemodialysis Single Group Assignment: All enrolled subjects will be connected to the CM-1500 for monitoring during their hemodialysis session
  CM-1500: The CM-1500 is a U.S. FDA cleared non-invasive monitoring device that simultaneously monitors five (5) parameters of a patient's body. A combination of these parameters is represented by a single number known as the Relative Index value.
Arm/Group | Hemodialysis Single Group Assignment
Number analyzed (Participants) | 15
Relative Index (RI) | 93.05 (0.43)

2. Secondary Outcome: Mean Intrasubject Variability (Standard Deviation) in Relative Index (RI) During Hemodialysis Sessions
Description: The secondary objective is to characterize intrasubject variability in RI changes across 3 hemodialysis sessions. Cohort intrasubject variability was calculated by averaging individual subject standard deviations across enrollments. Variability for each subject is calculated by finding the RI mean and standard deviation for all RI values (1 per sec) during all 3 monitoring sessions. The RI is an investigational value which utilizes proprietary algorithms to combine the changes of multiple measured parameters (utilizing a weighted summation of percent change values) which are indicative of relative changes in fluid volume in adult patients into a single value. The RI is a unitless value with no set min. or max. where 100 is a patient's baseline. Based on the nature of the RI itself, a direct interpretation of a positive or negative outcome cannot be derived from the absolute value, instead it could be used to monitor trending of a patient's parameters relative to their baseline.
Time Frame: Duration of standard dialysis procedure (Range: 131 to 241 minutes)
Population: Each subject was monitored for 3 separate hemodialysis sessions. Intrasubject variability was determined by comparing the 3 sessions for each subject against each other.
Measure: Mean (Standard Deviation); unit: Relative Index (RI)
Arm/Group | Hemodialysis Single Group Assignment
Number analyzed (Participants) | 15
Relative Index (RI) | 2.27 (2.07)

3. Secondary Outcome: Mean Intersubject Variability (Standard Deviation) in Relative Index (RI) During Hemodialysis Sessions
Description: The secondary objective is to characterize intersubject variability in RI changes across 3 hemodialysis sessions. Intersubject variability was calculated by finding the mean and standard deviation of the variability (standard deviation) from the mean RI values (1 value per sec) for each hemodialysis session monitoring period (3 sessions x 15 subjects = 45 individual monitoring sessions). The RI is an investigational value which utilizes proprietary algorithms to combine the changes of multiple measured parameters (utilizing a weighted summation of percent change values) which are indicative of relative changes in fluid volume in adult patients into a single value. The RI is a unitless value with no set min. or max., where 100 is a patient's baseline. Based on the nature of the RI itself, a direct interpretation of a positive or negative outcome cannot be derived from the absolute value, instead it could be used to monitor trending of a patient's parameters relative to their baseline.
Time Frame: Duration of standard dialysis procedure (Range: 131 to 241 minutes)
Measure: Mean (Standard Deviation); unit: Relative Index (RI)
Arm/Group | Hemodialysis Single Group Assignment
Number analyzed (Participants) | 15
Relative Index (RI) | 2.91 (3.27)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during subject participation and for 48hrs following the completion of subject participation, up to 17 days.
Arm/Group | Hemodialysis Single Group Assignment
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemodialysis Single Group Assignment (N=15)
Minor Adverse Event (Skin and subcutaneous tissue disorders) | 1 (1) — Subject experienced minor skin irritation/redness after electrode removal. Symptoms resolved without treatment and was designated as Not Serious by the Investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT05125848/Prot_SAP_000.pdf